CLINICAL TRIAL: NCT06490848
Title: Comparing the Safety and Efficacy of Cerebral Angiography Using Trans-femoral Approach Versus Trans-radial Approach
Brief Title: Comparing the Safety and Efficacy of Cerebral TFA and TRA Methods
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Humain Baharvahdat, Associate Professor of Endovascular Neurosurgery, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4001116
Record Dates: First submitted 2023-10-17; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Angiography

STUDY DESIGN:
Intervention Model Description: In this study, all consecutive patients referred for diagnostic cerebral angiography at a large academic tertiary care medical center were randomly assigned to two groups: right radial access versus femoral access for diagnostic cerebral angiography.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Transradial approach group (Active Comparator): The diagnostic angiography was performed by radial approach.
  Interventions: Procedure: Diagnostic cerebral angiography
- Trasfemoral approach group (Active Comparator): The diagnostic angiography was performed by femoral approach.
  Interventions: Procedure: Diagnostic cerebral angiography

INTERVENTIONS:
Procedure: Diagnostic cerebral angiography — In transradial access, no preprocedural upper extremity collateral blood supply testing was completed. When the radial access is unsuccessful, it is shifted to ulnar or femoral access. All right arms were secured in the fully supine position to allow access to both radial and ulnar arteries. At the conclusion of radial access procedures, a TR band was applied to close the access. Neurological exams as well as radial artery pulse and pulse oximeter of the right first finger were assessed during and on discharge by trained recovery nurses. Femoral access was performed in a standard manner. After the access (femoral or radial), a cerebral angiogram was performed in a standard manner using appropriate catheters (vertebral, bern, Simmons 2 or 3) according to the access. For the radial access, the patient was slightly sedated.

SUMMARY:
Transradial diagnostic angiography in cardiovascular disease given lower vascular complications. However, neuroendovascular surgeons have not widely adopted the transradial approach for diagnostic approach and interventional procedures. This study aims to compare the efficacy, safety, and patient satisfaction with the transradial approach versus the transfemoral approach in diagnostic cerebral angiography.

DETAILED DESCRIPTION:
Transradial diagnostic angiography in cardiovascular disease given lower vascular complications. However, neuroendovascular surgeons have not widely adopted the transradial approach for diagnostic approach and interventional procedures. This study aims to compare the efficacy, safety, and patient satisfaction with the transradial approach versus the transfemoral approach in diagnostic cerebral angiography.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive adult inpatients and outpatients referred for diagnostic cerebral angiography
* the presence of the right radial pulse and at least one femoral pulse

Exclusion Criteria:

* age<18
* pregnant patients
* occlusion of aorta or proximal both iliac/ femoral artery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
technical success | during procedure
  Incidence of sucess of performing the programmed cerebral angiogram through the randomised access without for crossover.
access success | during procedure
  Incidence of puncture success to insert a sheat in the access point

SECONDARY OUTCOMES:
total procedure time | during procedure
  the duration (minutes) between the insertion of sheath and removal of sheath. fluoroscopy time, the need for performing 3D angiography, dose area product (DAP), total radiation dose, successful puncture (successful insertion of radial artery sheath and femoral artery sheath). Procedures that yielded angiograms with acceptable quality through the subclavian artery injection (with an inflated blood pressure cuff on the arm), in cases of failed vertebral artery cannulation, were also considered successful.
total fluoroscopy time | during procedure
  the duration of fluoroscopy
complication | during procedure or one week after procedure
  incidence of any procedural-related complication procedure

OTHER OUTCOMES:
Patient Satisfaction | immediately after procedure, one hour after the procedure
  The pain evaluation by the Visual analog score (VAS) by trained nurses and recorded as the scoring system (No pain: 0; Mild:1-3; Moderate:4-7; Severe:8-10).

CONTACTS AND LOCATIONS:
Locations (1):
- Mashhad university of medical sciences, Mashhad, Razavi Khorasan Province, Iran